CLINICAL TRIAL: NCT00968656
Title: Assessment of Cellular Proliferation in Tumors by Positron Emission Tomography (PET) Using [18F]ISO-1
Acronym: FISO PET/CT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Isotrace Technologies (Unknown)
Responsible Party: Principal Investigator, Farrokh Dehdashti, Professor of Radiology, Washington University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FISO 08-1010
Record Dates: First submitted 2009-08-28; First posted 2009-08-31 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Breast Cancer; Head and Neck Cancer; Diffuse Large B-cell Lymphoma
Keywords: Breast cancer; Head and Neck Cancer; Diffuse Large B-cell lymphoma; Cellular proliferation
MeSH Terms: conditions — Breast Neoplasms; Head and Neck Neoplasms; Lymphoma, Large B-Cell, Diffuse; Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: PET/CT — Patients receive F-18-ISO-1 i.v. and undergo PET/CT imaging at 2-3 time points following the injection.
Other: Laboratory Testing — Blood and urine samples for laboratory analysis and radioactive counts will be obtained during the imaging sessions
Other: Safety Testing — ECG tracings, and vital signs (blood pressure, heart rate, body temperature and respiration rate) are obtained at several time points before, during, and after the imaging sessions.
Other: Immunohistochemistry staining — If available tissue from a biopsy or surgery will be tested cellular proliferation markers such as Ki67 and sigma 2 receptors
Drug: F-18-ISO — Patients receive F-18-ISO-1 i.v.

SUMMARY:
The main purpose of this study is to see if Positron Emission Tomography (PET) imaging with a radioactive tracer called 18F-ISO-1 can accurately identify how quickly cancer cells are growing or dividing. A second purpose for this study is to determine, by taking pictures, what tissues and organs of the body take up 18F-ISO-1 naturally and to determine how that uptake changes over time.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older with biopsy-proven breast cancer, head & neck cancer or diffuse large B-cell lymphoma.
* For determination of Ki-67, S-phase, mitotic index, and sigma-2 receptor assessment, cancer subjects must be scheduled to undergo surgical resection of the primary tumor without intervening therapy, or be scheduled to undergo (or have already undergone) tissue sampling as either standard of care or part of another research project prior to any planned treatment for their cancer. For tumor sigma-2 receptors assessment, about 0.5 g of fresh tumor tissue kept frozen on dry ice is needed, other proliferative markers may be determined on a much smaller specimen. Thus, it is possible that the analysis of sigma-2 receptors may not be possible in all patients, as obtaining 0.5 g tumor specimen may not practical in all patients.
* Newly diagnosed breast cancer, head & neck cancer, or diffuse large B-cell lymphoma subjects should have a primary lesion size ≥ 1.5 cm as determined by imaging studies (ultrasonography, mammography, CT or MRI) or physical examination and who have not received any treatment for their cancer.
* Able to give informed consent.
* Not currently pregnant or nursing: Female subjects must be either surgically sterile (has had a documented bilateral oophorectomy and/or documented hysterectomy), or post menopausal (cessation of menses for more than 1 year). If of childbearing potential, a urine pregnancy test must be performed within the 24 hour period immediately prior to administration of [18F]ISO-1 and determined to be negative.

Exclusion Criteria:

* Patients with other invasive malignancies, with the exception of non-melanoma skin cancer, who had (or have) any evidence of the other cancer present within the last 5 years. Lymphoma patients who have received treatment in the past but have a new diagnosis of diffuse large B-cell lymphoma are eligible to participate providing they will undergo tissue sampling as specified in the inclusion criteria.
* Unable to tolerate 60-90 minutes of PET imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
The primary out come is to assess the diagnostic quality of [18F]ISO-1-PET/CT images at the proposed 8 mCi dose. | 3 years

SECONDARY OUTCOMES:
Secondary outcome is to quantitatively determine the relationship between tumor [18F]ISO-1 uptake and Ki-67, S-phase, mitotic index and sigma-2 receptors content of the tumor. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Farrokh Dehdashti, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University / Barnes Jewish Hospital, St Louis, Missouri, United States